CLINICAL TRIAL: NCT05156177
Title: Correlation of Fecal Microbiome and Its Metabolites With Outcome of Radiotherapy in Locoregionally Advanced Head and Neck Squamous Cell Carcinoma (COMRAD-HNSCC)
Brief Title: Correlation of Fecal Microbiome and Its Metabolites With Outcome of Radiotherapy in Head and Neck Carcinoma
Acronym: COMRAD-HNSCC
Status: Active, not recruiting | Type: Observational
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Principal Investigator, Gaber Plavc, Principal Investigator, Institute of Oncology Ljubljana
Other Study IDs: ERIDEK-0052/2021
Record Dates: First submitted 2021-11-14; First posted 2021-12-14 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Radiotherapy; Microbiome; Metabolites
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preclinical studies have shown that the response of solid tumors and normal tissues to radiotherapy can be regulated by gut microbiota and its metabolites. In this study, the composition of gut microbiota in patients with locally advanced head and neck cancers undergoing definitive radiotherapy will be analysed together with bacterial metabolites in stool and blood and a possible correlation with treatment outcome and treatment toxicity will be determined.

DETAILED DESCRIPTION:
Head and neck cancer patients commonly present with unresectable locoregionally advanced disease in which radiotherapy is the mainstay of curative-intent treatment albeit at the cost of substantial acute and late toxicity. Recently discovered mechanisms by which gut microbiota and its metabolites impact tumor's and normal tissue's response to radiotherapy offer new ways to improve the therapeutic index of radiotherapy in solid tumors.

COMRAD-HNSCC is a prospective study assessing the correlation between gut microbiota composition and its metabolites and the response to radiotherapy in patients with unresectable locoregionally advanced head and neck cancer. Stool and serum samples will be collected at the beginning and at the end of curative radiotherapy treatment. The composition of gut microbiota will be analysed by ribosomal DNA high-throughput amplicon sequencing of the DNA isolated from stool samples, whereas targeted metabolomics using liquid chromatography-mass spectrometry will be performed on stool and serum samples.

The long-term goal of this study is to deepen the understanding of the role of gut microbiome and its metabolites in efficacy and toxicity of radiotherapy in head and neck cancer, and provide a basis for subsequent exploration to increase therapeutic index by regulating gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Signed written and voluntary informed consent.
* Patient must be willing and able to provide collection for stool specimen analyses at 2 time points.
* Age > 18 years, male or female.
* Patient must be diagnosed with histologically confirmed squamous cell carcinoma of the head and neck (oral cavity, oropharynx, larynx, hypopharynx, or nasopharynx).
* Patients must be eligible for curative-intent treatment with either radiotherapy or concurrent chemo-radiotherapy.
* Overall disease stage III-IV based on 8th edition of American Joint Committee on Cancer staging system.

Exclusion Criteria:

* Receipt of induction chemotherapy.
* Presence of distant metastases.
* Any previous head and neck cancer.
* Any other known concurrent malignant disease.
* Any condition that, in the opinion of the Investigator, would interfere with patient safety, or evaluation of the collected specimen and interpretation of study result.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects diagnosed with locoregionally-advanced head and neck squamous cell carcinoma being treated with definitive radiotherapy with or without concurrent chemotherapy at the Institute of Oncology Ljubljana.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 3 months post-treatment
  Objective response rate to radiotherapy according to RECIST 1.1 criteria as measured with computed tomography.
  Associations with differences in fecal microbiota composition and in bacterial metabolites will be made between responders and non-responders.
Acute radiation induced mucositis and dermatitis | Up to 3 months post-treatment
  Acute radiation induced mucositis and dermatitis according to CTCAE v3.0 as measured with clinical examination.
  Associations with differences in fecal microbiota composition and in bacterial metabolites will be made between patients with a maximum Grade ≤ 2 versus those with a maximum Grade > 3 acute radiation induced mucositis and dermatitis.

CONTACTS AND LOCATIONS:
Overall Officials: Gaber Plavc, MD, Principal Investigator — Institute of Oncology Ljubljana
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia